CLINICAL TRIAL: NCT07404319
Title: Randomised Control Trial of Effectiveness of Exercise Alone and tDCS+Exercise on Cognitive Function Improvement in Patients With Treatment Resistant Schizophrenia
Brief Title: Effectiveness of Exercise Alone and tDCS+Exercise on Cognitive Function Improvement in Patients With Treatment Resistant Schizophrenia
Acronym: TRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kit Wa Chan (Other)
Responsible Party: Sponsor-Investigator, Kit Wa Chan, Clinical Associate Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: C7001-24Y
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Schizophrenia; Treatment Resistant Schizophrenia; Cognitive Impairment
Keywords: tDCS; aerobic exercise; cognitive function; treatment-resistant schizophrenia
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Treatment-Resistant; Cognitive Dysfunction | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1: Aerobic Exercise + Active tDCS (Experimental): * Intervention 1 (Behavioral): Aerobic exercise
  * Intervention 2 (Device): Active tDCS
  Interventions: Behavioral: Aerobic Exercise; Device: Active tDCS
- Arm 2: Aerobic Exercise + Sham tDCS (Active Comparator): * Intervention 1 (Behavioral): Aerobic exercise
  * Intervention 2 (Device): Sham tDCS
  Interventions: Behavioral: Aerobic Exercise; Device: Sham tDCS
- Arm 3: Stretching/Education + Active tDCS (Active Comparator): * Intervention 1 (Behavioral): Stretching/education control
  * Intervention 2 (Device): Active tDCS
  Interventions: Behavioral: Stretching/Education Control; Device: Active tDCS
- Arm 4: Stretching/Education + Sham tDCS (Sham Comparator): * Intervention 1 (Behavioral): Stretching/education control
  * Intervention 2 (Device): Sham tDCS
  Interventions: Behavioral: Stretching/Education Control; Device: Sham tDCS

INTERVENTIONS:
Behavioral: Aerobic Exercise — * Dose: 18 sessions over 6 weeks (3/week)
  * Session duration: 45-60 minutes including warm up/cool down
  * Intensity: Moderate (target 60-75% HRR or RPE 12-15)
  * Mode: Aerobic dance
  * Delivery: Supervised by qualified staff; HR/RPE logged each session
  * Rationale: Exercise improves global cognition and domains such as working memory and attention/vigilance in schizophrenia; supervision/dose relate to effect size.
  Arms: Arm 1: Aerobic Exercise + Active tDCS; Arm 2: Aerobic Exercise + Sham tDCS
Behavioral: Stretching/Education Control — * Dose: 18 sessions over 6 weeks (3/week)
  * Session duration: 45-60 minutes
  * Intensity: Low (HR <40% HRR; RPE <10)
  * Components: Stretching + standardized health education modules
  * Purpose: Attention matched control to reduce contact/expectancy bias in non pharmacological trials.
  Arms: Arm 3: Stretching/Education + Active tDCS; Arm 4: Stretching/Education + Sham tDCS
Device: Active tDCS — * Montage: Anode F3 (left DLPFC), cathode Fp2 (right supraorbital)
  * Intensity: 2.0 mA
  * Duration: 20 minutes (30 s ramp up/down)
  * Schedule: 18 sessions (one per visit)
  * Rationale: Frontal tDCS protocols have shown promise for cognitive deficits and working memory in schizophrenia
  Arms: Arm 1: Aerobic Exercise + Active tDCS; Arm 3: Stretching/Education + Active tDCS
Device: Sham tDCS — • Same montage; ramp up then off (device standard sham) to mimic cutaneous sensations.
  Arms: Arm 2: Aerobic Exercise + Sham tDCS; Arm 4: Stretching/Education + Sham tDCS

SUMMARY:
Cognitive impairment is a major determinant of disability in schizophrenia. Aerobic exercise improves global cognition in schizophrenia, particularly working memory and attention/vigilance. Transcranial direct current stimulation (tDCS) targeting frontal regions has shown promise for cognitive deficits, including working memory improvements in some studies. This randomized 2×2 factorial trial will test the independent and combined effects of supervised aerobic exercise and prefrontal tDCS on cognition in treatment resistant schizophrenia, measured using the MATRICS Consensus Cognitive Battery (MCCB).

DETAILED DESCRIPTION:
This is an individually randomized, sham controlled (tDCS), assessor blinded 2×2 factorial clinical trial comparing: (1) aerobic exercise vs stretching/education control and (2) active vs sham prefrontal tDCS. The factorial design enables estimation of the main effects of exercise and tDCS and their interaction (synergy/antagonism) in one trial.

Participants with treatment resistant schizophrenia (TRS) will complete 18 sessions over 6 weeks (3 sessions/week). Each session includes tDCS (active or sham) during the physical activity condition (aerobic exercise or stretching/education) to standardize timing and contact. Evidence suggests exercise associated cognitive gains relate to intervention dose and supervision. Noninvasive brain stimulation outcomes may vary with stimulation dose parameters, supporting a standardized protocol.

Cognition will be assessed using the MCCB, which evaluates seven cognitive domains relevant to schizophrenia and yields an Overall Composite T score. The primary endpoint is Week 6 (end of intervention), with durability assessed at 3 months post intervention (Week 18).

ELIGIBILITY:
Inclusion Criteria:

* DSM 5 schizophrenia-spectrum disorders
* Treatment resistant schizophrenia: inadequate response to ≥2 antipsychotics of adequate dose/duration
* Clinically stable ≥4 weeks
* Able to provide informed consent

Exclusion Criteria:

* Neurological disorder (e.g., epilepsy, stroke) or significant head injury
* Implanted electronic devices / contraindications to tDCS; scalp lesions at electrode sites
* Medical contraindications to moderate aerobic exercise
* Substance dependence within 3 months (except nicotine)
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
MCCB Overall Composite T score change from baseline (Week 0) to end of intervention (Week 6). | 6 weeks
  MCCB provides standardized domain and composite T scores for schizophrenia cognition research.

SECONDARY OUTCOMES:
MCCB Working Memory Domain change (LNS + WMS III Spatial Span domain T score) baseline to Week 6. | 6 weeks
  Working memory is responsive to exercise in schizophrenia meta-analysis and frequently targeted in frontal tDCS studies.
MCCB Attention/Vigilance Domain change (CPT IP domain T score) baseline to Week 6. | 6 weeks
  Attention/vigilance improves with exercise in schizophrenia meta analysis; attention demanding performance may improve in some tDCS protocols.
Changes of negative symptoms measured with SANS from baseline to week 6 | 6 weeks
  Studies have shown effectiveness of exercise and tDCS on improvement of negative symptoms in patients with schizophrenia
Durability of changes of negative symptoms relative to baseline and week 6 | 18 weeks
  Evaluates the persistence of the improvement of negative symptoms

OTHER OUTCOMES:
Durability: MCCB Overall Composite and key domains at 3 months post intervention (Week 18) relative to baseline and Week 6. | 18 weeks total
  Evaluates persistence of cognitive gains.
Changes of social functioning measured with SOFAS from baseline to 18 weeks | 18 weeks
  Cognitive function and negative symptoms are closely related to social functioning. Improvement of these may contribute to the improvement of overall social functioning
Durability: MCCB Overall Composite and key domains at 6 months post intervention (Week 24) relative to baseline and Week 6 and week 18 | 24
  Evaluates persistence of cognitive gains
Durability of improvement of negative symptoms at 6 months after intervention (week 24) relative to baseline, week 6 and week 18 | 24 weeks
  Evaluates persistence of the improvement of negative symptoms
Durability of the improvement of social functioning at 6 months post intervention (week 24) relative to baseline and week 18 | 24 weeks
  Evaluates the persistence or even further improvement of the social functioning

CONTACTS AND LOCATIONS:
Overall Officials: Kit Wa Chan, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Sharing data will depend on funder. Further information will need to be checked and confirmed.